CLINICAL TRIAL: NCT01658254
Title: A Cohort Randomized Controlled Trial Evaluating the Effect of Sending a Reminder to Responsible Parties of Clinical Trials in the Posting of Basic Results Onto ClinicalTrials.Gov
Brief Title: Posting of Basic Results of Clinical Trials
Acronym: REGIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PR 738
Record Dates: First submitted 2012-06-20; First posted 2012-08-06 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2012-06

CONDITIONS: The Study Will Focus on no Specific Conditions
Keywords: Clinical trials; Basic results; Registry

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Survey by email (Experimental): One arm of investigators will receive the survey to answer by email, reminding the necessity of posting basic results
  Interventions: Other: survey by email
- Non interventional arm (No Intervention): This arm will receive no intervention (no email with the survey)

INTERVENTIONS:
Other: survey by email — The intervention consists in an email to be sent to the sponsor and/or principal investigator of randomly assigned trials. This email will notify them that their trial's primary completion date is over a year old and will ask the reasons why they have not posted results on the registry. Several reasons will be proposed, and investigators or sponsors will be asked to reply by sending back an email or through a website where the same questions will appear. A follow-up email will systematically be sent 7 days after, with similar content (appendix2). The emails will be sent as direct emails, without attached files, with the edit subject "Posting basic results". The controlled group will receive no intervention.
  Arms: Survey by email

SUMMARY:
The gap between the high number of registered trials and the few ones where results were available (in registries or in journals) has been identified as a major problem distorting the scientific evidence available. As a consequence, the FDAAA (Food and Drug Administration Amendments Act) added on September 27, 2007 a requirements policy regarding publication of summary results on the publicly accessible registry ClinicalTrials.gov. Reporting of summary results is required for "applicable clinical trials" no later than one year after the "primary completion date", i.e. the date of collection of primary outcome data on the last patient to be enrolled. 'Applicable clinical trials', is the term used in the FDAAA to designate trials that may be subject to the registration and reporting requirements.

Not complying with the reporting requirements can result in penalties, such as withholding of National Institute of Health grant or funding and civil monetary penalties of up to $10,000 a day. Despite the possibility of incurring penalties for not complying with the posting requirement, compliance remains globally poor.

In this current study, the primary objective will be to test the hypothesis that sending an email looking as a survey, reminding the necessity of posting results to the trials' responsible parties registered in ClinicalTrials.gov and subject to mandatory reporting but not complying with it, will increase the results posting rate.

DETAILED DESCRIPTION:
According to the recommendation of 2005 by International Committee of Medical Journal Editors (ICMJE), clinical trials must be registered before enrolment of the first patient in a free registry recognized by the World Health Organization (WHO). The goal is to improve transparency of clinical research. The ClinicalTrials.gov trial registry, initiated subsequently to the US Food and Drug Administration Modernization Act (FDAMA) in 1997, is the widest used registry, and contains more than 121 000 studies located in 179 countries (data of March 1, 2012).

The gap between the high number of registered trials and the few ones where results were available (in registries or in journals) has been identified as a major problem distorting the scientific evidence available, and inducing publication bias. As a consequence, the FDAAA (Food and Drug Administration Amendments Act) added on September 27, 2007 a requirements policy regarding publication of summary results on the publicly accessible registry ClinicalTrials.gov. Reporting of summary results is required for "applicable clinical trials" no later than one year after the "primary completion date", i.e. the date of collection of primary outcome data on the last patient to be enrolled. 'Applicable clinical trials', is the term used in the FDAAA to designate trials that may be subject to the registration and reporting requirements. They include interventional controlled studies registered after the enactment of the FDAAA (or ongoing at this date), involving drugs, biologics, or devices (only after FDA-approved for any use), regardless of sponsorship; phases II through IV; located at least in one U.S. site.

The entity or individual responsible for registering and posting basic results is called the 'responsible party'. This term refers to the sponsor of the study or the principal investigator of the study, if so designated by a sponsor, grantee, contractor, or awardee.

In certain circumstances, delayed submission of results information with certification can be allowed. Not complying with the reporting requirements can result in penalties, such as withholding of National Institute of Health grant or funding and civil monetary penalties of up to $10,000 a day. Despite the possibility of incurring penalties for not complying with the posting requirement, compliance remains globally poor.

In this current study, the primary objective will be to test the hypothesis that sending an email asking to answer a survey, reminding the necessity of posting results to the trials' responsible parties registered in ClinicalTrials.gov and subject to mandatory reporting but not complying with it, will increase the results posting rate.

The secondary objective will be to investigate the reasons given by the trials' responsible parties for not posting summary results onto the registry.

ELIGIBILITY:
Inclusion Criteria:

* Interventional studies of drugs, biological or devices
* Studies which are closed and either completed or active but not recruiting anymore
* Studies with at least one site in the USA
* Studies registered as phase IV
* Studies with a primary completion date or, if missing, a completion date ranging from October 2008 to January 2011
* Studies without posted results on the registry

Exclusion Criteria:

* Studies which are still recruiting
* Studies which are either withdrawn or suspended
* Studies which primary completion date is less than one year
* Studies without a given primary completion date or completion date
* Studies involving interventions which are neither drugs or biologics nor devices will be excluded
* Studies whose summary results are posted
* Studies without indication on the sponsor or the principal investigator
* Studies whom email address of the sponsor or the principal investigator could not be found in a publicly accessible site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The proportions of trials with posted results at 90 days will be compared using a chi-square test to the control group. | 90 days
  Primary endpoint: the proportions of trials with posted results on the registry at 90 days will be compared to the control group using a chi-square test.

SECONDARY OUTCOMES:
The proportions of trials with posted results on the registry at 180 days will be compared to the control group using a chi-square test. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Ravaud, MD, PhD, Principal Investigator — Hotel-Dieu, Clinical Epidemiology Center
Locations (1):
- Clinical Epidemiology Center, Hotel-Dieu, Paris, France

REFERENCES:
- [Derived] Maruani A, Boutron I, Baron G, Ravaud P. Impact of sending email reminders of the legal requirement for posting results on ClinicalTrials.gov: cohort embedded pragmatic randomized controlled trial. BMJ. 2014 Sep 19;349:g5579. doi: 10.1136/bmj.g5579. PMID 25239625